CLINICAL TRIAL: NCT01527214
Title: The Effect of Direct Referral for Fast CT Scan in Early Lung Cancer Detection in General Practice. Clinical, Randomised Trial
Brief Title: The Effect of Direct Referral for Fast CT Scan in Early Lung Cancer Detection in General Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DirectCT
Record Dates: First submitted 2012-01-20; First posted 2012-02-06 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Lung Cancer
Keywords: Lung cancer; early detection; CT scan; General Practice; Effect of Computed Tomography scans; Clinical medical education
MeSH Terms: conditions — Lung Neoplasms | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT scan and education (Experimental): All general practices referring to the Department of Pulmonary Medicine, Aarhus University Hospital.Randomized 1:1. In the intervention group, GPs continue to refer to the lung cancer fast track when indicated. In addition, they are allowed to refer directly to a rapid chest CT scan in cases where they find reasons to examine the patient for lung diseases without having sufficient suspicion of lung cancer to refer the patient to the lung cancer fast track. The GPs will be offered special training related to the diagnosis of lung cancer in general practice before the new referral option is introduced. This will be done by offering training sessions and written material.
  Interventions: Radiation: CT scan and education
- Control (No Intervention): Cluster eligibility: all practices referring to the Department of Pulmonary Medicine, Aarhus University Hospital. Randomized 1:1. Control arm continues with the usual referral pattern

INTERVENTIONS:
Radiation: CT scan and education — GPs get direct access to chest CT scans for their patients. The GPs will be offered special training related to the diagnosis of lung cancer in general practice.This will be done by offering training sessions and written material. The training will include risk groups, alarm symptoms, symptom complexes and interpretation of CT scan descriptions.
  Arms: CT scan and education

SUMMARY:
Background: The primary investigation of lung cancer (LC) is for 85% of the cases conducted through General Practice, sadly it tends to take a relatively long time from first time the patient is seen by their General Practitioner and until they are diagnosed. LC symptoms are common, but usual because of benign diseases. Only 33% of LC patients presenting with alarm symptoms. On average a General Practitioner in Denmark sees only one patient with newly diagnosed lung cancer a year and the doctor will therefore get the clinical experience that when they refer a patient, test often come out negative and they therefore fail to refer and delay will increase - with a poorer prognosis as a result. Centrally in the diagnosis is conventional chest X-ray, which unfortunately is inefficient in many cases, while CT scanning has proven effective even for small tumors.

Hypothesis and aims: The project has three main hypotheses to be tested 1) the GP's use of cancer fast-track and detection of suspected lung cancer can be optimized in relation to interpretation of symptoms and subsequent referral practices and radiological investigation. 2) General Practitioners with special training can change the referral routines and 3) direct access to fast CT scanning leads to earlier diagnosis of lung cancer.

Methods: The first part of the study is a register-based study of lung cancer patients' road to diagnosis, based on a database of newly diagnosed cancer patients in a year. Second part of the study is a clinical, randomized study of the effect of referral directly to fast chest CT scan. Primary endpoint is delay, secondary endpoints are referral pattern (use of fast-track packet), primary use of CT and 1-year mortality. Furthermore side effects, including patient groups with increased delay.

The study will contribute new knowledge to the way GP's interpret symptoms, the way they refer their patients when they suspect cancer, their use of diagnostic imaging and cancer fast-track pathways. It will then provide a unique opportunity to create the necessary knowledge about the effects of direct referral to fast CT scan and it might be a decision aid whether to open for direct CT scan in General Practice for a group of patients.

ELIGIBILITY:
Inclusion Criteria:

* all practices referring to the Department of Pulmonary Medicine, Aarhus University Hospital.

Exclusion Criteria:

* former lung cancer patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Delay | 12 month
  Time from first presentation i General Practice to the patient obtains the diagnosis

SECONDARY OUTCOMES:
Referral pattern (use of fast-track packet) | 12 month
Primary use of CT | 12 month
1-year mortality. | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vedsted, Professor, Principal Investigator — The Research Unit for Generel Practice
Locations (1):
- University of Aarhus, Aarhus, Aarhus, Denmark

REFERENCES:
- [Derived] Guldbrandt LM, Fenger-Gron M, Rasmussen TR, Rasmussen F, Meldgaard P, Vedsted P. The effect of direct access to CT scan in early lung cancer detection: an unblinded, cluster-randomised trial. BMC Cancer. 2015 Nov 25;15:934. doi: 10.1186/s12885-015-1941-2. PMID 26608727
- [Derived] Guldbrandt LM, Rasmussen TR, Rasmussen F, Vedsted P. Implementing direct access to low-dose computed tomography in general practice--method, adaption and outcome. PLoS One. 2014 Nov 10;9(11):e112162. doi: 10.1371/journal.pone.0112162. eCollection 2014. PMID 25383780